CLINICAL TRIAL: NCT03626922
Title: A Phase IB Study of Pembrolizumab in Combination With Pemetrexed and Oxaliplatin in Patients With Chemo-Refractory Metastatic Colorectal Cancer
Brief Title: Study of Pembrolizumab With Pemetrexed and Oxaliplatin in Chemo-Refractory Metastatic Colorectal Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-10
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: NSABP; Merck & Co; Eli Lilly and Company; Pembrolizumab; Pemetrexed; Oxaliplatin; MSS mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Pemetrexed; Oxaliplatin; Dexamethasone; Calcium Dobesilate; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Pembrolizumab + Pemetrexed every 21 days. Folic Acid 5 days prior to first dose of pemetrexed and daily including 21 days after last dose of pemetrexed.
  Dexamethasone twice daily on the day before, the day of, and the day after each dose of pemetrexed.
  Vitamin B-12 7 days prior to first dose of pemetrexed, every 9 weeks, continue until 3 weeks after last dose of pemetrexed.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Dexamethasone; Dietary Supplement: Folic Acid; Dietary Supplement: Vitamin B-12
- Cohort 2 (Experimental): Pembrolizumab + Pemetrexed + Oxaliplatin every 21 days. Folic Acid 5 days prior to first dose of pemetrexed and daily including 21 days after last dose of pemetrexed.
  Dexamethasone twice daily on the day before, the day of, and the day after each dose of pemetrexed.
  Vitamin B-12 7 days prior to first dose of pemetrexed, every 9 weeks, continue until 3 weeks after last dose of pemetrexed.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Oxaliplatin; Drug: Dexamethasone; Dietary Supplement: Folic Acid; Dietary Supplement: Vitamin B-12

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV on Day 1 of each 21 day cycle until maximum of 35 cycles.
  Other Names: Keytruda
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV on Day 1 of each 21 day cycle until maximum of 35 cycles.
  Other Names: Alimta
Drug: Oxaliplatin — Oxaliplatin-Dose level1: 85 mg/m2 IV on Day 1 of each 21 day cycle until a maximum of 35 cycles or until discontinued due to patient election, toxicity, disease progression.
  Dose level 2: 120 mg/m2 IV on Day 1 of each 21 day cycle until a maximum of 35 cycles or until discontinued due to patient election, toxicity, disease progression.
  The MTD dose of oxaliplatin in the study combination of Cohort 2 will be the recommended Phase II dose (RP2D) for the cohort expansion.
  Other Names: Eloxatin
  Arms: Cohort 2
Drug: Dexamethasone — Dexamethasone-4 mg by mouth twice daily on: the day before, the day of, and the day after each dose of pemetrexed.
  Other Names: Ozurdex
Dietary Supplement: Folic Acid — Folic Acid-400 micrograms by mouth daily starting 5 days prior to first dose of pemetrexed and continue daily to include 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B-12 — 1000 micrograms administered intramuscularly 7 days prior to the first dose of pemetrexed, every 9 weeks, and should continue until 3 weeks after the last dose of pemetrexed.

SUMMARY:
This is a Phase Ib study to evaluate the safety and preliminary anti-tumor activity of pembrolizumab in combination with pemetrexed with or without oxaliplatin in patients with chemo-refractory microsatellite stable (MSS) metastatic colorectal cancer (mCRC) without any further standard treatment options.

DETAILED DESCRIPTION:
The co-primary endpoints of the study are to 1) establish the recommended Phase II dose (RP2D) of pembrolizumab in combination with pemetrexed and oxaliplatin and 2) evaluate the antitumor efficacy.

The secondary aims of the study are to 1) evaluate the clinical benefit rate (CBR) of pembrolizumab in combination with pemetrexed and with pembrolizumab in combination with pemetrexed and oxaliplatin in patients with chemo-refractory MSS mCRC and 2) to estimate the progression free survival (PFS) and 3) overall survival (OS) in patients with MSS mCRC treated with pembrolizumab and pemetrexed or with pembrolizumab in combination with pemetrexed and oxaliplatin.

Patients enrolled to Cohort 1 will receive: pembrolizumab 200mg IV and pemetrexed 500 mg/m2 on Day 1 of each 21 day cycle.

Cohort 2 (the dose escalation portion of the study) will be a standard "3+3" design; 2 dose levels are planned. The first 3 to 6 patients in cohort 2 will be treated at dose level 1 and will receive pembrolizumab 200 mg IV, pemetrexed 500 mg/m2 IV and oxaliplatin 85 mg/ m2 on Day 1 of each 21 day cycle. If 1 of 3 patients in this cohort experiences a dose-limiting toxicity (DLT), see Section 6.4, 3 more patients will be added at the same dose level. If 0 of 3 initial patients or 1 of 6 patients in the cohort experiences a DLT, the dose for the next cohort will be escalated to dose level 2 and will receive pembrolizumab 200 mg IV, pemetrexed 500 mg/m2 IV and oxaliplatin 120 mg/ m2 on Day 1 of each 21 day cycle; otherwise, the combination will be considered too toxic. If ≥ 2 DLTs are experienced at any dose level, the combination will be considered too toxic and the next lower dose level will be considered the RP2D. A total of 12 patients will be treated at the RP2D as the expansion portion.

Patients in both cohorts will continue to receive study therapy (maximum of 35 cycles) unless therapy is discontinued due to patient election, toxicity, or disease progression.

Dose limiting toxicity (DLT) will be monitored during the first 21 days (Cycle 1) of each dose level in Cohort 2 and will be used for purposes of dose escalation and determination of RP2D. A DLT is defined as a non-hematologic adverse event (AE) of grade ≥ 3 or a hematologic toxicity of grade ≥ 4. Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0.

The highest dose level tolerable without dose limiting toxicities (DLTs) in < 2 of 6 patients will be considered the recommended phase 2 dose (RP2D) and be expanded to 12 patients.

The maximum total enrollment of the study is 33 patients. In Cohort 1, a total of 15 patients with chemo-refractory MSS mCRC will be treated for further safety assessment and a preliminary signal. In Cohort 2, 3 to 6 patients will be accrued per dose level. A total of 12 patients with chemo-refractory MSS mCRC will be treated on the RP2D for further safety and preliminary efficacy signal. Cohort 1 and Cohort 2 will be analyzed separately.

Efficacy will be evaluated as the individual best overall response as defined by a modified RECIST 1.1 (mRECIST 1.1). The objective response rate (complete response [CR] and partial response [PR]) will be determined. In either dose level cohort > 3 patients (> 3 of 18) with objective response (PR or CR) will warrant further investigation.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and, prior to beginning specific study procedures, must have signed and dated an appropriate IRB-approved consent form that conforms to federal and institutional guidelines for study treatment.
* The ECOG performance status must be 0 or 1.
* There must be histologic or cytologic confirmation of a diagnosis of microsatellite stable (MSS) colorectal adenocarcinoma using CLIA certified IHC or PCR-based MSI testing.
* Metastatic or locally advanced disease not amenable to curative surgery and/or radiotherapy.
* There must be documentation by PET/CT scan, CT scan, or MRI that the patient has evidence of measurable metastatic disease per RECIST 1.1.
* Patients must have had prior treatment for metastatic or unresectable for cure of colorectal cancer with standard chemotherapy including fluoropyrimidine-, oxaliplatin- and irinotecan- based chemotherapy, and if RAS wild-type, an anti-EGFR therapy.
* At the time of study entry, blood counts performed within 2 weeks prior to study entry must meet the following criteria:

  * ANC must be greater than or equal to 1500/mm3;
  * Platelet count must be greater than or equal to 100,000/mm3; and
  * Hemoglobin must be greater than or equal to 9 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 2 weeks prior to study entry must be met:

  * Total bilirubin must be less than or equal to 1.5 x ULN.
  * AST and ALT must be less than or equal to 2.5 x ULN for the lab except in the presence of known hepatic metastasis, wherein transaminases may be up to 5 x ULN.
  * Alkaline phosphatase must be less than or equal to 3 x ULN for the lab.
* International normalized ratio of prothrombin time must be less than or equal to 1.5 times the ULN. Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no underlying abnormality in coagulation parameters exists per medical history. For laboratories that do not report an ULN for the INR assay, use less than or equal to 1.2 as the value for the ULN.
* Creatinine must be less than or equal to 1.5 x upper limit of normal (ULN) and measured or calculated creatinine clearance (CrCl) greater than or equal to 60mL/min.
* All hematologic, gastrointestinal, and genitourinary chemotherapy toxicities must be less than grade 2 at the time study therapy is to begin. (Note: Transfusions may be used to correct hemoglobin for patients experiencing anemia from therapy who otherwise would be eligible for the study.
* Patients must be able to interrupt nonsteroidal anti-inflammatory drugs (NSAIDS) 2 days before (5 days for long acting NSAIDS), the day of and 2 days following administration of pemetrexed.
* Patients must be able to take folic acid, vitamin B12, and dexamethasone per protocol.
* Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Male and female patients with reproductive potential must agree to use accepted effective methods of contraception while receiving study therapy and for at least 120 days after the completion of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

* Diagnosis of anal or small bowel carcinoma.
* Colorectal cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy.
* Use and/or receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal anti-bodies) or radiation therapy within 4 weeks prior to receiving first dose of study therapy.
* Prior monoclonal antibody therapy within 4 weeks prior to first dose of FC-10 study therapy or who has not recovered (i.e., less than or equal to grade 1 or at baseline) from adverse events due to a previously administered agent.
* Neuropathy greater than grade 1.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. Note: steroid use is permitted only as indicated per protocol.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study therapy. Administration of killed vaccines is allowed.
* Known history of hepatitis B or hepatitis C.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment.
* Active infection or chronic infection requiring systemic therapy.
* Known history of human immunodeficiency virus (HIV) or acquired immunodeficiency-related (AIDS) illnesses.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) is not allowed.
* History of allogeneic organ transplantation.
* Any of the following cardiac conditions:

  * Documented NYHA Class III or IV congestive heart failure,
  * Myocardial infarction within 6 months prior to study entry,
  * Unstable angina within 6 months prior to study entry,
  * Symptomatic arrhythmia.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Ongoing or active gastritis or peptic ulcer disease.
* Presence of third space fluid which cannot be controlled by drainage. Active bleeding diatheses.
* Known history of previous diagnosis of tuberculosis.
* History of hypersensitivity to pembrolizumab, pemetrexed, or oxaliplatin or any excipients of these drugs.
* Known history or confirmation of active pneumonia, non-infectious pneumonitis that requires steroids, current pneumonitis, symptomatic interstitial lung disease, or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization.
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, and basal cell and squamous cell carcinoma of the skin.
* Psychiatric or addictive disorders or other conditions that in the opinion of the investigator would preclude the patient from meeting the study requirements or interfere with interpretation of study results.
* Pregnancy or lactation at the time of study entry.
* Use of any investigational agent within 4 weeks prior to the first dose study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate to pembrolizumab plus pemetrexed | From initiation of pembrolizumab and pemetrexed until disease progression, intolerable toxicity, or completion of 35 cycles (each cycle is 21 days), approximately 2 years.
  Objective Response Rate using modified RECIST 1.1.
Objective Response Rate to pembrolizumab and pemetrexed plus oxaliplatin | From initiation of pembrolizumab and pemetrexed plus oxaliplatin until disease progression intolerable toxicity, or completion of 35 cycles (each cycle is 21 days), approximately 2 years.
  Objective Response Rate using modified RECIST 1.1.

SECONDARY OUTCOMES:
Frequency of Adverse Events | From begining of study therapy until disease progression, intolerable toxicity, or completion of 35 cycles (each cycle is 21 days), approximately 2 years.
  Frequency of adverse events in Cohort 1 categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0.
Frequency of Adverse Events | From begining of study therapy until disease progression, intolerable toxicity, or completion of 35 cycles (each cycle is 21 days), approximately 2 years.
  Frequency of adverse events in Cohort 2 categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0.
Clinical Benefit Rate | From initiation of study therapy until disease progression, approximately 2 years.
  Rate of disease status by continuous tumor measurement using modified RECIST 1.1.
Progression-Free Survival | From initiation of study therapy until disease progression, approximately 2 years.
  Progression-free survival (PFS). Percentage of patients alive with absence of progression assessed using RECIST 1.1 criteria.
Overall Survival | Time of study entry through 1 year.
  Overall Survival. Percentage of patients alive after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (15):
- United States (15):
  - UF Health Davis Cancer Pavilion & Shands Medical Plaza, Gainesville, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cancer Care Specialists of Central IL-Swansea, Swansea, Illinois
  - University of Michigan-Oncology, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan-Brighton Center for Specialty Care, Brighton, Michigan
  - Minnesota Oncology-Minneapolis, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - HealthPartners Riverside Clinic, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium-MMCORC, Saint Louis Park, Minnesota
  - Thomas Jefferson University Hospital-Sidney Kimmel Cancer Network, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania